CLINICAL TRIAL: NCT05055752
Title: A Randomized, Actively-Controlled, Crossover Bioequivalence Study of a Novel Pharmaceutical Lipid-Aspirin Complex Formulation at 325 mg Dose Versus Immediate Release Aspirin in Healthy Volunteers
Brief Title: Randomized, Crossover Bioequivalence Study of PL-ASA Versus Immediate Release Aspirin in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PL-ASA-009
Record Dates: First submitted 2021-09-16; First posted 2021-09-24 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-09

CONDITIONS: Bioequivalence

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, single dose 2-way crossover study in healthy volunteers
Who Masked: Outcomes Assessor
Masking Description: All investigators, Sponsor personnel, clinical monitors, independent PK analyst, and subjects in the study will be unblinded to the treatment allocation as all of the primary and secondary endpoints are based on objective criteria of laboratory findings. Laboratory personnel involved in the analysis will be blinded to the treatment allocation
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PL-ASA capsule, then IR-ASA tablet (Other): One PL-ASA 325 mg capsule, 14 day washout then one IR-ASA 325 mg tablet
  Interventions: Drug: Pharmaceutical-lipid aspirin (PL-ASA)
- IR-ASA tablet, then PL-ASA capsule (Other): One IR-ASA 325 mg tablet, 14 day washout, then one PL-ASA 325 mg capsule,
  Interventions: Drug: Pharmaceutical-lipid aspirin (PL-ASA)

INTERVENTIONS:
Drug: Pharmaceutical-lipid aspirin (PL-ASA) — Subjects receive the first drug, followed by a 7-day washout period, then receive the second drug.
  Other Names: Immediate-release aspirin (IR-ASA)

SUMMARY:
This trial is a randomized, actively-controlled, open-label, 2-way crossover bioequivalence study to determine PK parameters following treatment with test aspirin product (PL-ASA capsules) and reference aspirin product (IR-ASA tablets) administered at a single dose of 325 mg.

DETAILED DESCRIPTION:
Healthy volunteers will be asked to sign informed consent prior to conduct any protocol specified activities at screening. A total of 20 eligible subjects will be randomized, in a fasted state, to 1 of 2 sequences of study drug administration (each study drug dose contains 325 mg aspirin) at 1:1 ratio:

* PL-ASA capsule, IR-ASA tablet
* IR-ASA tablet, PL-ASA capsule

After completion of the first treatment on Day 1 and following the 24 hours of sample collection, a minimum of a 7-day washout period will be required before all subjects are crossed over and receive treatment with the alternative compound; i.e., subject randomized to receive PL-ASA capsule as a first treatment will receive IR-ASA tablet as the second treatment, and vice-versa.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age without known acute or chronic medical conditions requiring treatment;
* If female, a negative pregnancy test and not nursing;
* If female and of childbearing potential, use of adequate birth control for the duration of the study (i.e., barrier methods such as female diaphragm or male condom; intrauterine devices, hormonal implants, pill, patch, shot, vaginal ring, etc.; total abstinence from heterosexual intercourse when it is in line with the preferred and usual lifestyle of the subject; vasectomized partner);
* Non-smoker, including no use of any smoking cessation nicotine-containing products (i.e., nicotine replacement therapy [patch, spray, inhaler, gum, lozenge, bupropion SR, clonidine and nortriptyline], e-cigarettes, etc.) for at least 3 months prior to screening;
* Consumes on average no more than 2 alcoholic drinks (1 drink is defined as approximately 12 oz of regular beer, 5 oz of wine, or 1.5 oz of hard liquor) per day for at least 30 days prior to screening;
* A body mass index (BMI) between 18 to 32 kg/m2;
* Agrees to refrain from alcohol consumption for 48 hours prior to and 48 hours after drug administration; and
* Able and willing to provide written informed consent prior to the study.

Exclusion Criteria:

* Abnormal screening/baseline laboratory parameters deemed to be clinically significant by the Investigator;
* Positive urine alcohol and drug screen result;
* Use of any prescription medications other than hormone replacement therapy, thyroid replacement therapy, or oral contraceptive within 3 days prior to study drug administration;
* Use of antacid medications, including over-the-counter (OTC) products within 3 days prior to study drug administration;
* Use of dietary or herbal supplements containing salicylates, fish oil, or any vitamins within 2 weeks of study drug administration;
* Use of any of the following medications within 2 weeks prior to study drug administration:

  1. Non-steroidal anti-inflammatory drugs (NSAIDs), including aspirin or aspirin-containing products and acetaminophen.
  2. Any anti-platelet agent, including clopidogrel, prasugrel, ticagrelor, ticlopidine, cangrelor, dipyridamole, cilostazol, vorapaxar, abciximab, eptifibatide, tirofiban, or triflusal.
  3. Any anti-coagulant agent, including warfarin, acenocoumarol, phenprocoumon, phenindione, rivaroxaban, dabigatran, apixaban, edoxaban, heparin, enoxaparin, fondaparinux, ximelagatran, argatroban, lepirudin, hirudin, or bivalirudin.
* Use of an investigational agent within the past 30 days prior to drug administration.
* Hypersensitivity or contraindications to aspirin, ibuprofen, or other NSAID;
* Soy allergy or sensitivity;
* History of:

  1. Gastrointestinal problems including ulcers, frequent indigestion, or frequent heartburn.
  2. Coronary disease, stroke, or congestive heart failure.
  3. Asthma, nasal polyps, or angioedema other than resolved childhood asthma.
  4. Kidney or liver disease.
  5. Thrombocytopenia, neutropenia, bleeding disorder, or history of non-trauma related hemorrhage.
  6. Chronic hypertension.
* Current enrollment in another investigational trial; or
* History of cancer within the last 5 years (except for skin cancer resolved by excision, or cervical cancer adequately treated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of single-dose acetylsalicylic acid PK of the PL-ASA formulation to IR-ASA in healthy volunteers at 325 mg dose level. | 24 hours after dosing
  Bioequivalence using serum determinations of acetylsalicylic acid concentration

CONTACTS AND LOCATIONS:
Locations (1):
- PRA-EDS, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No